CLINICAL TRIAL: NCT03133312
Title: A Single Site Prospective Randomized Controlled Trial Comparing Chlorhexidine Gluconate and Povidone-Iodine as Vaginal Preparation Antiseptics for Cesarean Section to Determine Effect on Bacterial Load
Brief Title: Chlorhexidine Gluconate Versus Povidone-Iodine as Vaginal Preparation Antiseptics Prior to Cesarean Delivery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Metro Health, Michigan (Other)
Responsible Party: Principal Investigator, Brad Irving, DO, FACOOG, Principal Investigator, Metro Health, Michigan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: VAGPrep
Record Dates: First submitted 2017-04-03; First posted 2017-04-28 (Actual); Last update posted 2019-03-11 (Actual); Status verified 2019-03

CONDITIONS: Infection, Bacterial
MeSH Terms: conditions — Bacterial Infections | interventions — chlorhexidine gluconate; Paint; Povidone-Iodine

STUDY DESIGN:
Intervention Model Description: Drug: Chlorhexidine Gluconate Applied to vagina pre-operatively for antiseptic; regulated as a drug by FDA
  Other Name: CHG
  Drug: Povidone-Iodine Scrub and Paint Applied to vagina pre-operatively for antiseptic; regulated as a drug by FDA
  Other Name: Betadine
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participant will not know which group they have been assigned to. The surgeon and OR staff performing the vaginal preparation will know, but the nursing staff in the recovery area will not. The lab will be blinded toward which type of surgical prep was used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Chlorhexidine Gluconate (Experimental): Pre-operative vagina preparation with Chlorhexidine Gluconate Intervention: Drug: Chlorhexidine Gluconate Other Name: Chlora-Prep
  Interventions: Drug: Chlorhexidine Gluconate
- Povidone-Iodine Scrub and Paint (Experimental): Pre-operative vagina preparation with Povidone-Iodine Scrub and Paint Intervention: Drug: Povidone-Iodine Scrub and Paint Other Name: Betadine
  Interventions: Drug: Povidone-Iodine Scrub and Paint

INTERVENTIONS:
Drug: Chlorhexidine Gluconate — Pre-operative vaginal preparation with 4% Chlorhexidine Gluconate Intervention
  Other Names: Chlora-Prep
  Arms: Chlorhexidine Gluconate
Drug: Povidone-Iodine Scrub and Paint — Pre-operative vaginal preparation with 10% Povidone-Iodine Scrub and Paint Intervention
  Other Names: Betadine
  Arms: Povidone-Iodine Scrub and Paint

SUMMARY:
Primary Hypothesis: chlorhexidine gluconate antiseptic vaginal preparation is superior to povidone-iodine vaginal preparation in decreasing the bacterial load within the vagina when prepping prior to a cesarean section.

DETAILED DESCRIPTION:
Patients who are planning cesarean will be recruited and consented for study participation at time of admission to labor and delivery.

Patients undergoing cesarean who meet inclusion/exclusion criteria will be randomized to one of two surgical preparations as follows: 1. Chlorhexidine gluconate (CHG); or, 2. Povidone-iodine scrub. Randomization will be performed by the consenting surgeon (listed as key personnel) after the patient has arrived into the operating room for cesarean. To establish baseline bacterial load, a qualitative BAL culture will be collected prior to the vaginal preparations. Pre-operative surgical site antisepsis will be performed according to randomization. All other surgical practices will remain at the surgeon's discretion according to standard of care at Metro Health Hospital.

At the completion of the cesarean, it is standard practice to perform a manual evacuation of blood clots from the lower uterine segment. The study culture will be obtained by the consenting surgeon immediately prior to manual evacuation. The cultures will then be sent to the lab for determination of total bacterial load of the vaginal area. The lab will be blinded toward which type of vaginal prep was used. Total colony count will be determined by certified lab personnel by adding all counts regardless of bacteria type. A secondary chart review will be performed by the investigator within 30 days of the postoperative period to evaluate for length of hospital stay, pain level, blood loss, any additional antibiotics received postoperatively, and the development of post-operative infection in subjects up to 30 days after discharge.

The research project will take place over a 12-month period of time at Metro Health Hospital. In review of Metro Health Labor and Delivery statistics for scheduled cesarean sections performed in 2016, an average of 18.8 were performed a month, giving a total of approximately 226 in a one-year period. Based on the research study published by Culligan, Kubik, Murphy, et al. comparing the two vaginal preparations for vaginal hysterectomy, an estimated sample size was calculated. Using the 90 minute colony counts of 20,472 (40,058) vs 1,221 (2,857), and using an alpha of .05 and power of 80% investigator found the sample size for each group should be at least 27. This sample size (27 X 2 groups) is very close to the sample size (50) in the Culligan experiment. In an attempt to ensure the most clinically significant, investigators anticipate screening between 70-100 patients with approximately 70-80% participation.

Analysis will be performed by the investigators for completeness, accuracy, strict adherence to study protocol, safety, and statistical significance. The investigators are also subject to periodic audits by the Institutional Review Board (IRB).

ELIGIBILITY:
Inclusion Criteria:

* Scheduled low transverse cesarean section (can be primary or repeat)
* Term gestation ≥ 37 weeks

Exclusion Criteria:

* Allergy to either antiseptic
* Rupture of amniotic membranes
* Preterm gestation
* Active labor
* Emergency or unscheduled cesarean sections
* Infection diagnosis on admission
* Vaginal infection or any treatment of vulvovaginitis in prior 7 days
* Patients under the age of 18 years

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 100 (Actual)
Dates: Start 2017-05-02 (Actual); Primary Completion 2017-12-30 (Actual); Study Completion 2017-12-30 (Actual)

PRIMARY OUTCOMES:
Bacterial Load | Immediately Post-operative prior to exit from operating room
  Change in total bacterial load from baseline (pre-operative) vaginal culture

SECONDARY OUTCOMES:
Length of Hospital Stay | 2 or 3 post-operative days
  Number of days

OTHER OUTCOMES:
Post-Operative Infection | up to 30 day post-operative
  Presence of post-operative infection including endometritis, pelvic abscess, and skin/wound

CONTACTS AND LOCATIONS:
Overall Officials: Brad Irving, DO, FACOOG, Principal Investigator — Metro Health
Locations (1):
- Metro Health, Wyoming, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Culligan PJ, Kubik K, Murphy M, Blackwell L, Snyder J. A randomized trial that compared povidone iodine and chlorhexidine as antiseptics for vaginal hysterectomy. Am J Obstet Gynecol. 2005 Feb;192(2):422-5. doi: 10.1016/j.ajog.2004.08.010. PMID 15695981
- [Result] Darouiche RO, Wall MJ Jr, Itani KM, Otterson MF, Webb AL, Carrick MM, Miller HJ, Awad SS, Crosby CT, Mosier MC, Alsharif A, Berger DH. Chlorhexidine-Alcohol versus Povidone-Iodine for Surgical-Site Antisepsis. N Engl J Med. 2010 Jan 7;362(1):18-26. doi: 10.1056/NEJMoa0810988. PMID 20054046
- [Result] Levin I, Amer-Alshiek J, Avni A, Lessing JB, Satel A, Almog B. Chlorhexidine and alcohol versus povidone-iodine for antisepsis in gynecological surgery. J Womens Health (Larchmt). 2011 Mar;20(3):321-4. doi: 10.1089/jwh.2010.2391. Epub 2011 Feb 16. PMID 21323582
- [Result] Tuuli MG, Liu J, Stout MJ, Martin S, Cahill AG, Odibo AO, Colditz GA, Macones GA. A Randomized Trial Comparing Skin Antiseptic Agents at Cesarean Delivery. N Engl J Med. 2016 Feb 18;374(7):647-55. doi: 10.1056/NEJMoa1511048. Epub 2016 Feb 4. PMID 26844840
- [Derived] Haas DM, Morgan S, Contreras K, Kimball S. Vaginal preparation with antiseptic solution before cesarean section for preventing postoperative infections. Cochrane Database Syst Rev. 2020 Apr 26;4(4):CD007892. doi: 10.1002/14651858.CD007892.pub7. PMID 32335895